CLINICAL TRIAL: NCT05320861
Title: A Single Dose Study Designed to Assess the Mass Balance Recovery, Absorption, Metabolism and Excretion of [14C]SJP-0008 in Healthy Male Subjects After an Oral Dose
Brief Title: Single Dose ADME Study of [14C]SJP-0008 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Senju Pharmaceutical Co., Ltd. (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJP-0008/1-02; 2021-002615-65 (EudraCT Number); 18pc0101026h0001 (Other Grant/Funding Number: The Japan Agency for Medical Research and Development)
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: Mass Balance Recovery; Metabolite Profile; Metabolite Identification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]SJP-0008 (Experimental)
  Interventions: Drug: [14C]SJP-0008

INTERVENTIONS:
Drug: [14C]SJP-0008 — Single oral dose of [14C]SJP-0008

SUMMARY:
This single centre, open-label, non-randomised, single period, single-dose study in healthy male subjects was designed and conducted to assess the mass balance recovery, PK, metabolite profile and metabolite identification of SJP-0008.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
* Must be willing and able to communicate and participate in the whole study
* Must have regular bowel movements
* Must provide written informed consent
* Must agree to adhere to the contraception requirements of the protocol

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Subjects who are, or are immediate family members of, a study site or sponsor employee
* Subjects who report to have previously received SJP-0008
* Evidence of current SARS-CoV-2 infection
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 6 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 6 months
* Subjects with pregnant or lactating partners
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study

Other protocol-defined exclusion criteria may apply

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity in all excreta after a single oral dose of [14C]SJP-0008 | Until the mass balance criteria for all participants have been met (estimated up to Day 10)
  Mass balance recovery of total radioactivity in all excreta by analysing the total radioactivity and metabolic profile in plasma, urine and faeces samples.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of SJP-0008 and SNJ-2026 | Up to Day 8
Area under the concentration-time curve from time zero to last measurable concentration (AUC0-last) of SJP-0008 and SNJ-2026 | Up to Day 8
Area under concentration-time curve from time zero to infinity (AUC0-inf) of SJP-0008 and SNJ-2026 | Up to Day 8
Area under the concentration-time curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUCextrap) of SJP-0008 and SNJ-2026 | Up to Day 8
Time to maximum plasma concentration (Tmax) of SJP-0008 and SNJ-2026 | Up to Day 8
Half-life (T1/2) of SJP-0008 and SNJ-2026 | Up to Day 8
First order rate constant associated with the terminal (log-linear) portion of the curve (Lambda-z) of SJP-0008 and SNJ-2026 | Up to Day 8
Percentage of participants with adverse events (AEs) | Until the mass balance criteria for all participants have been met (estimated up to Day 10)

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No